CLINICAL TRIAL: NCT01943760
Title: Evaluation of the Analgesic Effect of Tramadol Wound Infiltration in Children Under Inguinal Hernioplasty. A Double-blind, Randomized Study.
Brief Title: Tamadol Wound Infiltration in Children Under Inguinal Hernioplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Laura Albertoni Giraldes, doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 187177
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Children; Inguinal Hernia
Keywords: Tramadol; Children; Hernioplasty; Wound infiltration
MeSH Terms: conditions — Hernia, Inguinal | interventions — Tramadol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tramadol wound infiltration (Active Comparator): 2 mg / kg of tramadol diluted in 5 ml of 0.9% saline solution wound infiltration 20ml of 0.9% saline solution intravenously
  Interventions: Drug: tramadol; Drug: 0.9% saline
- tramadol intravenous administration (Experimental): 2 mg / kg of tramadol diluted 20ml of 0.9% saline solution intravenously 5 ml of 0.9% saline solution wound infiltration
  Interventions: Drug: tramadol; Drug: 0.9% saline

INTERVENTIONS:
Drug: tramadol — The volume of the solution was adequate to maintain the concentration of 2% tramadol
  Other Names: tramal
Drug: 0.9% saline

SUMMARY:
Tramadol is a centrally acting analgesic, is primarily Indicated for the treatment of acute pain, moderate to severe. The hernioplasty in children is an outpatient procedure, and the possibility of postoperative analgesia with fewer systemic adverse effects such as nausea and vomiting make the tramadol infiltration a technique of interest. There is controversy about its effectiveness.

The local effect of tramadol in hernioplasty was also studied by researchers with some better postoperative analgesia than with local anestetic .

There are few studies with administration of tramadol for hernioplasty, Which led to the interest in this study.

DETAILED DESCRIPTION:
The primary objective of the study was to evaluate the analgesic effect of tramadol injected into the surgical incision in patients undergoing hernioplasty.

The study is a prospective, comparative, double covered. The distribution of patients in the groups was randomly drawn prior to starting the project and the groups were identified in envelopes numbered 1-40.

Criteria for inclusion and exclusion After approval by the Ethics Committee of UNIFESP and signature of consent by those responsible, and the term of assent by patients over six years, 40 children of both sexes will be evaluated, aged between 3 and 12 years who underwent hernioplasty.

Children with bleeding disorders, using analgesic or sensitivity to any drug will be excluded.

The patients will be randomly divided into one of two groups. Patients in group 1 will receive local infiltration with 2 mg / kg of tramadol diluted in 5 ml of 0.9% saline solution and 20ml of 0.9% saline solution intravenously at the end of the surgical procedure Patients in group 2 will receive 2 mg.kg-1 tramadol intravenously diluted in 20 ml of 0.9% saline solution and local infiltration with 5 mL of saline solution 0.9% at the end of the surgical procedure.

All patients will undergo general anesthesia, and will receive additional analgesia with dipyrone and morphine as needed in post operative period.

ELIGIBILITY:
Inclusion Criteria:

* children of both sexes
* aged between 3 and 12 years
* underwent hernioplasty

Exclusion Criteria:

* children with bleeding disorders
* using analgesic
* sensitivity to any drug.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity after wound infiltration with tramadol | 1 month
  Faces scale

CONTACTS AND LOCATIONS:
Overall Officials: Ana LA Giraldes, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- São Paulo Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Demiraran Y, Ilce Z, Kocaman B, Bozkurt P. Does tramadol wound infiltration offer an advantage over bupivacaine for postoperative analgesia in children following herniotomy? Paediatr Anaesth. 2006 Oct;16(10):1047-50. doi: 10.1111/j.1460-9592.2006.01910.x. PMID 16972834